CLINICAL TRIAL: NCT02578394
Title: A Feasibility Study to Undertake a Definitive Randomised Multi-centre, Double-blind, Double-dummy Controlled Study of a Novel Agent Anakinra vs. Depo-Medrone for Acute Gout Attacks in Patients With Moderate Chronic Kidney Disease
Brief Title: Anakinra vs. Steroids for the Treatment of Gout Attacks in Patients With Renal Disease (ASGARD): A Feasibility Study
Acronym: ASGARD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other); University of East Anglia (Other); University of Essex (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P0850; 2015-001787-19 (EudraCT Number); PB-PG-0614-34090 (Other Grant/Funding Number: National Institute of Health Research)
Record Dates: First submitted 2015-10-02; First posted 2015-10-19 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Gout; Chronic Kidney Diseases
Keywords: Gout; Kidney; Depo-Medrone; Anakinra
MeSH Terms: conditions — Gout; Renal Insufficiency, Chronic | interventions — Interleukin 1 Receptor Antagonist Protein; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Anakinra 100mg and Placebo Depo-Medrone
  Interventions: Drug: Anakinra 100mg and Placebo Depo-Medrone
- Group B (Active Comparator): Depo-Medrone 120mg and Placebo (Anakinra)
  Interventions: Drug: Depo-Medrone 120mg and Placebo (Anakinra)

INTERVENTIONS:
Drug: Anakinra 100mg and Placebo Depo-Medrone — Anakinra 100mg injection S/C Day 1 to Day 5 and Placebo Depo-Medrone (Lipofundin 3mL) I/M Day 1. Anakinra is an interleukin-1 receptor antagonist. Placebo for Depo-Medrone placebo is Lipofundin MCT/LCT 10%.
  Other Names: Kineret
  Arms: Group A
Drug: Depo-Medrone 120mg and Placebo (Anakinra) — Depo-Medrone 120mg in 3mL. Placebo for Anakinra supplied from manufacturer. 120mg Depo-Medrone I/M Day 1 and Placebo Anakinra 100mg injection S/C Day 1 to Day 5.
  Other Names: Methylprednisolone Acetate
  Arms: Group B

SUMMARY:
The aim of this study is to determine the feasibility of running a phase III double-blind, double-dummy randomised controlled trial comparing Depo-Medrone 120mg intramuscular injection vs. Anakinra 100mg subcutaneous injection for 5 days for the treatment of acute gout attacks in patients with chronic kidney disease as defined by a eGFR < 60mls/min/1.73m2 and ≥ 30mls/min/1.73m2.

DETAILED DESCRIPTION:
Gout is a common condition that affects 1 in 40 people in the UK. It causes painful "attacks" of joint swelling, redness and tenderness, mostly affecting the foot, ankle, knee, hand and wrist. It is common in people with kidney disease, who also tend to be older people with other medical conditions such as high blood pressure, heart disease and diabetes. The investigators do not know the safest and best way to treat gout attacks in this increasing cohort of people. A lot of people are given treatment that can worsen their kidney disease, along with their other medical conditions.

The investigators want to compare the safest treatment currently available, steroids, with a new treatment called Anakinra. This treatment stops the action of a chemical called interleukin-1 which has been discovered to play an important role in gout attacks. This treatment has already been used to treat gout attacks in a handful of patients with kidney disease. The investigators feel it may be a better alternative to steroid treatment which can sometime worsen diabetes, heart disease and blood pressure. Participants will predominantly be followed-up for one week and a final 8 week follow-up, and be recruited from hospitals in the East of England.

A definitive scientific study comparing these two treatments would involve a big expensive study requiring large numbers of patients and large amounts of information to be collected. Before the investigators do a big study like this, the investigators want to perform a small study using a smaller number of patients (32 patients) over a period of 22 months in total. It will then give us information to plan a larger study to answer the question of which treatment may be better, safer and provides the most value for money for the NHS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects capable of giving informed consent.
2. Male or non-pregnant, non-nursing female
3. ≥ 18 years of age
4. eGFR < 60mls/min/1.73m2 and ≥ 30mls/min/1.73m2 as calculated using serum creatinine and modified MDRD formula as per renal association guidelines.
5. Diagnosis of gout arthritis as defined by the American College of Rheumatology 1977 preliminary criteria (this criteria is currently endorsed by NICE guidelines).
6. Gout flare less ≤ 36 hours
7. Baseline pain intensity > or equal to 50mm on the 0-100 mm VAS. In the case of multiple joints (≤ 3), the most affected joint will be assessed.

Exclusion Criteria:

1. Treatment with NSAIDS in last 48 hours, systemic steroids in last 4 weeks or colchicine within 7 days.
2. Polyarticular gout, i.e. affecting four or more 4 joints
3. Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis such as systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis.
4. Con-current immunosuppression/immunomodulatory treatment (Calcineurin inhibitor, anti-proliferative or biologic) therapy for other reason i.e. organ transplant.
5. Prior history or current inflammatory joint disease other than gout (e.g. rheumatoid arthritis (RA), reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease). Concurrent medication for RA like methotrexate and anti-TNF treatment has been associated with increased risk of neutropenia and infection.
6. Current active malignancy (with the exception of basal cell or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia and non-metastatic/advanced prostate cancer).
7. Any patients with contra-indication to intramuscular injection such as coagulopathy or thrombocytopenia (Platelet count<100 x 109/L (100,000/mm3)).
8. Abnormal liver function tests: Total bilirubin>upper limit of normal, Alanine aminotransferase (ALT) or Aspartate Aminotransferase (AST) >2 times upper limit of normal.
9. Haemoglobin <85g/L (8.5 g/dL)
10. White blood cell (WBC) count<1.5 x 109/L (1000/mm3), absolute neutrophil count<1.5 x 109/L (1000/mm3)
11. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), hepatic, endocrine (including uncontrolled diabetes) or gastrointestinal disease.
12. Known positive hepatitis B virus surface antigen (HBsAg), hepatitis C (HCV) antibody or HIV.
13. Females of child bearing potential who are not willing to use highly effective birth control methods from the time of consent to one week after treatment discontinuation. Highly effective method of contraception (hormonal or barrier method of birth control; abstinence) consist of:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; oral, intravaginal, transdermal.
    * Progestogen-only hormonal contraception associated with inhibition of ovulation; oral, injectable, implantable.
    * Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion or vasectomised partner
    * Sexual abstinence
14. Females of childbearing potential must have a negative pregnancy test (highly sensitive urine or serum pregnancy test after a confirmed menstrual period) within 7 days prior to treatment initiation. Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
15. Females must not be breastfeeding.
16. Patients who have had treatment as part of this trial cannot have repeat treatment for another flare as part of the trial.
17. Patient with allergies to excipients of IMPs: citric acid, anhydrous, sodium chloride, disodium edetate dehydrate, polysorbate 80, sodium hydroxide. Hypersensitivity to E. Coli derived proteins, egg proteins and soy proteins. Patients with a latex allergy are also not eligible as the inner needle cover of the pre-filled syringe contains dry natural rubber (a derivative of latex).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Resolution of pain: time to 50% reduction and complete resolution of pain in self-assessed pain intensity in the joint most affected. | Baseline (Day 1) to Day 7
  VAS (0-100mm) and 5-point Likert scale.

SECONDARY OUTCOMES:
Participant reported outcome measure of treatment response | Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7
  5-point Likert scale score
Physician / Investigator assessment of joint tenderness and swelling | Day 1, Day 2, Day 4 and Day 7
  4-point Likert scale score
Participant assessment of activity limitation | Day 1, Day 2, Day 5, Day 7
  Lower Extremity Functional Scale score
Participant assessment of activity limitation and quality of life | Day 1, Day 2, Day 4, Day 7 and 8 weeks
  EQ-5D-5L health states will be used to calculate the index. Health profiles will be obtained and Quality Adjusted Life Years will be derived
Participant assessment of activity limitation and quality of life using HAQ-DI | Day 1, Day 7 and 8
  Scores calculated from single scales and each dimension
Participant assessment of quality of life | Day 1, Day 7 and 8
  SF-36 score
Healthcare resource use | 8 weeks
  Highly modified client service use inventory score
CRP | Day 1, Day 4 and Day 7
  Changes in CRP
White Cell Count | Day 1, Day 4 and Day 7
  Changes in white cell count. Number of participants who develop neutropenia
eGFR | Day 1, Day 4 and Day 7
  Changes in eGFR
Safety reporting | Day 1 to 8 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Gowrie Balasubramaniam, MB ChB, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (1):
- Southend Hospital, Southend-on-Sea, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balasubramaniam G, Parker T, Turner D, Parker M, Scales J, Harnett P, Harrison M, Ahmed K, Bhagat S, Marianayagam T, Pitzalis C, Mallen C, Roddy E, Almond M, Dasgupta B. Feasibility randomised multicentre, double-blind, double-dummy controlled trial of anakinra, an interleukin-1 receptor antagonist versus intramuscular methylprednisolone for acute gout attacks in patients with chronic kidney disease (ASGARD): protocol study. BMJ Open. 2017 Sep 5;7(9):e017121. doi: 10.1136/bmjopen-2017-017121. PMID 28877949